CLINICAL TRIAL: NCT06065956
Title: Comparison of Hemodynamic Changes With Morphine Versus Esmolol as an Adjuvant Agent During Induction of Anaesthesia
Brief Title: Comparison of Hemodynamic Changes With Morphine Versus Esmolol During Induction of Anaesthesia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pakistan Navy Station Shifa Hospital (Other)
Responsible Party: Principal Investigator, Kenan Anwar Khan, FCPS 2 Registrar in Anaesthesiology, Pakistan Navy Station Shifa Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 433/8/22
Record Dates: First submitted 2023-08-29; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Intubation Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine group (Experimental): Half of participants will be comprising of morphine group
  Interventions: Drug: Intravenous morphine
- Esmolol group (Experimental): Half of participants will be comprising of esmolol group
  Interventions: Drug: Intravenous morphine

INTERVENTIONS:
Drug: Intravenous morphine — Morphine group(an opioid), participants were given intravenous morphine(an opioid) at induction of General Anaesthesia before laryngoscopy and intubation.
  The other group,Esmolol group(cardioselective beta blocker), participants were given intravenous esmolol(cardioselective beta blocker) during induction of General Anesthesia before laryngoscopy and intubation.
  Other Names: Intravenous esmolol

SUMMARY:
Comparing hemodynamic changes with morphine versus esmolol as an adjuvant agent during induction of Anaesthesia

DETAILED DESCRIPTION:
Comparing hemodynamic profile of patients during induction of General Anesthesia with intravenous morphine as an adjuvant drug versus Intravenous esmolol as an adjuvant agent,My aim is to study which drug has superior hemodynamic profile in terms of hemodynamic stability of patient requiring General Anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA 2 patients presenting for elective surgery.

Exclusion Criteria:

* Patients having major cardiac disease.
* Metastatic disease.
* Pregnant females.
* Those unwilling to be part of study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 06 months
  Change in blood pressure between baseline value and post Intubation value will be measured in millimeter of mercury (mmHg).
Pulse rate | 06 months
  Change in pulse rate between baseline value and post intubation value will be measured per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- PNS Shifa Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No